CLINICAL TRIAL: NCT01742416
Title: Ultrasound Assisted Arterial Cannulation in Small Children - To See or Not to See?
Brief Title: Ultrasound Assisted Arterial Cannulation in Small Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Katherine Taylor, Staff Anesthesiologist, The Hospital for Sick Children
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1000030723
Record Dates: First submitted 2012-11-30; First posted 2012-12-05 (Estimated); Last update posted 2019-07-05 (Actual); Status verified 2019-07

CONDITIONS: Arterial Cannulation
Keywords: Arterial Cannulation; Ultrasound; Palpation Method; Pediatrics; Cardiac Surgery; Craniotomies; Cranial Vault Surgery; Abdominal Procedures
MeSH Terms: interventions — High-Energy Shock Waves

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ultrasound (Experimental)
  Interventions: Procedure: Ultrasound
- Palpation Method (Active Comparator)
  Interventions: Procedure: Palpation Method

INTERVENTIONS:
Procedure: Ultrasound — Arterial cannulation facilitated by ultrasound.
  Arms: Ultrasound
Procedure: Palpation Method — Arterial cannulation by palpation method.
  Arms: Palpation Method

SUMMARY:
Arterial cannulation is a commonly performed invasive procedure in the operation room, the emergency department, and in the intensive care unit. The indications include the need for continuous blood-pressure monitoring, frequent arterial blood-gas analysis, and repeated blood sampling for laboratory evaluation. This procedure can be challenging even in the best of hands. Traditionally, the artery is located by feeling the pulse of the patient. The pulse may, however be weak or absent in patients with hypotension, edema, obesity or local thrombosis due to previous arterial cannulation in the same location. Furthermore, the catheter may not be passed successfully into the artery, despite apparent good blood return on initial puncture, or hematoma and spasms of the artery may develop after failed attempts, thus making further attempts even more difficult. While ultrasound (US) is being used with increasing frequency for central venous access, fewer clinicians are familiar with US-guided arterial catheterization. The aim of this study is to investigate if ultrasound facilitates arterial cannulation in children ≤24 months compared with the palpation method and to investigate the potential extra costs/savings of introducing the method. This study hypothesizes that the ultrasound method will facilitate arterial cannulation in small children compared with the palpation method.

ELIGIBILITY:
Inclusion Criteria:

* Children 24 months or younger
* Children undergoing elective surgical procedures where arterial cannulation is planned by the attending anaesthetist. These procedures include cardiac surgery, craniotomies, cranial vault surgery, and some abdominal procedures.

Exclusion Criteria:

* Refusal of consent from the parents
* Refusal of participation from the anaesthetist
* Children with anticipated circulatory instability after anaesthesia induction

  1. Pulmonary hypertension defined as an estimated pulmonary arterial pressure which is greater than or equal to 66% of systemic blood pressure
  2. Children with severe heart failure (right and/or left)

Ages: 1 Day to 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2012-11; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Number of Attempts | Change from baseline to successful cannulation (estimated average of 30 minutes)
  To measure the number of attempts to cannulate the artery per participant.

SECONDARY OUTCOMES:
Time to Successful Cannulation | Change from baseline to successful cannulation (estimated average of 30 minutes)
  To measure the difference between the time when the palpating finger touches the skin (palpation group) or the gel is applied to the skin (US group) at the first intended cannulation site and the time when the arterial cannula is correctly in place.
Rate of Success of First Attempt | Change from baseline to success of first attempt, when artery is successfully cannulated on first attempt (estimated average of 30 minutes)
  The rate of success of first attempt to cannulate the artery of each participant.
Number of Attempted Sites | Change from baseline to successful cannulation (estimated average of 30 minutes)
  To measure the total number of attempted sites.
Learning Curve | At approximately 4 months
  To measure the learning curve for each of the participating anaesthetist.
Cost of Procedure | Duration of the study (6 months)
  To measure the estimated cost of the procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Katherine Taylor, MD, Principal Investigator — The Hospital for Sick Children
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada